CLINICAL TRIAL: NCT02743598
Title: Effects of Liraglutide on Cognition, Chronic Inflammation and Glycemic Control in Overweight and Obese, HIV-infected Subjects With Type 2 Diabetes.
Brief Title: Liraglutide for HIV-associated Neurocognitive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding and time
Sponsor: Temple University (Other)
Collaborators: The Comprehensive NeuroAIDS Center (CNAC) at Temple University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23284
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: HIV Infection; Diabetes Mellitus Type 2; Obesity; Overweight; Metabolic Syndrome
Keywords: HIV infection; Diabetes Mellitus type 2; Obesity; Neurocognitive function
MeSH Terms: conditions — HIV Infections; Diabetes Mellitus, Type 2; Obesity; Overweight; Metabolic Syndrome | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liraglutide (Experimental)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide

SUMMARY:
This study will test the effect of liraglutide on cognitive function in HIV-infected overweight or obese subjects with type 2 diabetes.

DETAILED DESCRIPTION:
HIV, insulin resistance and type 2 diabetes mellitus (DM) are independently associated with cognitive impairment. Considering the synergistic effects of HIV and DM on cognition, these subjects are at increased risk of cognitive impairment. glucagon-like peptide 1 (GLP-1) receptors have wide tissue distribution including the central nervous system. The study hypothesis is that GLP-1 could potentially ameliorate the impairments in cognition in this population. This study will assess the impact of liraglutide on neurocognitive performance and peripheral inflammatory markers. It will also evaluate the effects of liraglutide on glycemic control and metabolic risk factors in HIV infected subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HIV controlled on therapy for at least 12 weeks
* Viral load < 200 copies
* BMI >27 to 45
* Diagnosis of DM type 2 with A1-C >7 to 15
* Participants must be willing to comply with all study related procedures

Exclusion Criteria:

* Personal or family history of pancreatitis
* Medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia Syndrome Type 2 (MEN 2)
* Gastroparesis
* Allergy to liraglutide or any of the active ingredients in liraglutide or other GLP-1 analogue
* Weight loss drugs other than metformin
* Type 1 diabetes mellitus or diabetic ketoacidosis
* Known major cognitive deficit dementia, history of head trauma with loss of consciousness >30 min, history of stroke, current central nervous system (CNS) disorder such as seizures or opportunistic CNS infection
* Renal insufficiency defined as creatinine clearance < 60 mL/min
* Active opportunistic infections
* Pregnancy or breastfeeding
* Unstable cardiovascular disease with hospitalization within 1 year for acute coronary syndrome
* Decompensated heart failure
* Substance abuse
* Active alcohol or opioid substitution therapy
* Serious or unstable medical or psychological conditions that would compromise the subject's safety for successful participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Neurocognitive performance- change in global cognitive scores on a standard neuropsychological profile | 6 months
Neurocognitive performance- change in domain averages on a standard neuropsychological profile | 6 months

SECONDARY OUTCOMES:
Change from baseline high sensitivity C-reactive protein | 3 and 6 months
Change from baseline d-dimer | 3 and 6 months
Change from baseline Interleukin 6 | 3 and 6 months
Change from baseline plasma soluble cluster of differentiation 14 (CD14) | 3 and 6 months
Change from baseline BMI | 3 and 6 months
Change from baseline weight | 3 and 6 months
Change from baseline waist circumference | 3 and 6 months
Change from baseline blood pressure | 3 and 6 months
Change from baseline serum triglycerides | 3 and 6 months
Change from baseline insulin resistance by homeostasis model assessment (HOMA-IR) in subjects not on insulin | 3 and 6 months
Change from baseline liver enzymes aspartate aminotransferase and alanine aminotransferase | 3 and 6 months
Change from baseline Hemoglobin A1c | 3 and 6 months
Change from baseline fructosamine | 3 and 6 months
Number of Adverse events | 3 and 6 months
Number of subjects with Adverse events | 3 and 6 months
Change from baseline serum LDL | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Vaz, MD Dipl ABOM, Principal Investigator — Temple University
Locations (1):
- Cherie Vaz, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No